CLINICAL TRIAL: NCT02058797
Title: Efficacy of Coherence Therapy for Procrastination: a Randomized Controlled Trial
Brief Title: Efficacy of Coherence Therapy for Procrastination
Acronym: CTFORPRO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Coherence Therapy intervention could not be delivered in a reliable and valid way for a variety of reasons.
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTprocrast
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Procrastination
Keywords: Procrastination; Coherence Therapy; Cognitive Behavioral Therapy; Repertory Grid Technique; Cognitive Conflicts; Personal Dilemmas
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coherence Therapy (Experimental): Individual treatment with Coherence Therapy: three one-hour sessions + one booster session.
  Interventions: Behavioral: Coherence Therapy
- Cognitive Behavioral Therapy (Active Comparator): Individual treatment with Cognitive Behavioral Therapy: three one-hour sessions + one booster session.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Coherence Therapy — Manualized individual treatment (3 + 1 one-hour sessions)
  Arms: Coherence Therapy
Behavioral: Cognitive Behavioral Therapy — Manualized individual treatment (3 + 1 one-hour sessions)
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to determine the efficacy of Coherence Therapy in treating procrastination. For that, this intervention is compared to Cognitive-Behavioral Therapy which was already proved to be efficacious in treating this problem. The method used is a randomized controlled trial.

DETAILED DESCRIPTION:
Procrastination is a recognized difficulty that entails negative outcomes regarding performance and subjective well-being. In order to find effective treatments for procrastination, the present study wants to test the efficacy of Coherence Therapy, compared with Cognitive Behavioral Therapy. Procrastination, negative emotional states and cognitive structure will be assessed in pre-treatment and post-treatment evaluation. A total of 30 students will be randomly assigned to Coherence Therapy (n=15) or Cognitive Behavioral Therapy (n=15). In both forms of treatment students will receive three weekly sessions and one more session six to seven weeks after the third session. The treatment will be provided by trained psychotherapists. Findings would clarify the effectiveness of Coherence Therapy for the treatment of procrastination and the change of emotional states and cognitive structure of the students after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being a student
* 19-26 years old
* A score above 51 on the General Procrastination Scale

Exclusion Criteria:

* Being currently under a psychological treatment
* Being diagnosed lately with any mental disorder
* Mental retardation
* Substantial visual, hearing or cognitive deficits
* Psychotic symptoms
* Organic brain dysfunction

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
General Procrastination Scale (Lay, 1986) | Post-treatment assessment (10-12 weeks)
  Change from Baseline in General Procrastination Scale measured before and after the therapy in order to determine the level of general procrastination.

OTHER OUTCOMES:
Repertory Grid Technique (Kelly, 1995; adaptation of Feixas & Cornejo, 1996) | Post-treatment assessment (10-12 weeks)
  Change in cognitive structure measured by Kelly's Repertory Grid Technique.
Depression, Anxiety and Stress Scale (Lovibond & Lovibond, 1995) | Post-treatment assessment (10-12 weeks)
  Change from Baseline in negative emotional states on three dimensions: depression, anxiety and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, Ph.D., Principal Investigator — University of Barcelona
Locations (1):
- University of Barcelona, Barcelona, Catalonia, Spain